The New Internet Generation: iCBT Treatment for Seniors With Mild-moderate Depression - a Pragmatic Randomised Controlled Trial in the Primary Care Context

ID: iCBT-Senior-DEP-2024-PRCT

August 15, 2024

## Statistical analysis plan

Descriptive statistics will be employed to summarize the data. Continuous variables will be assessed using independent sample t-tests or Mann-Whitney U tests, depending on the distribution of the data. Categorical variables and frequencies will be analyzed with Pearson chi-square tests.

To evaluate the primary outcome of depressive symptoms and quality of life (QoL) scores, we will use mixed model analysis with repeated measures. This approach will allow us to compare intra-individual changes between the intervention and control groups over time. The models will be adjusted for age, sex, education, antidepressant use at baseline, and the response variable at baseline.

Statistical analyses will be performed using SPSS and SAS software. A p-value of less than 0.05 will be considered statistically significant.